CLINICAL TRIAL: NCT05716789
Title: The Success Rate of Cardiopulmonary Resuscitation in Sudden Cardiac Arrest
Brief Title: Cardiopulmonary Resuscitation in Cases of Sudden Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Osama Hamdy
Record Dates: First submitted 2023-01-28; First posted 2023-02-08 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Cardiac Arrest
Keywords: CPR; Success Rate; Emergency medicine; Critical care; ICU and Pain Management
MeSH Terms: conditions — Heart Arrest; Agnosia | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CPR asseement (Experimental): determine the success rate of CPR in Emergency room and factors predicting successful CPR
  Interventions: Procedure: CPR

INTERVENTIONS:
Procedure: CPR — CPR in cardiac arrest patients

SUMMARY:
Determination the success rate of CPR on adults in Emergency room and predicting the factors that makes CPR is successful.

DETAILED DESCRIPTION:
Cardiac arrest is a medical emergency that requires immediate cardiopulmonary resuscitation (CPR). Return of spontaneous circulation (ROSC) is a core outcome element of cardiopulmonary resuscitation (CPR) both in out-of-hospital cardiac arrest (OHCA) and in-hospital cardiac arrest and has been considered a standard in the evaluation of successful resuscitation.

ROSC was defined as a clinical assessment that shows signs of life comprising of a palpable pulse for at least 20 minutes or generating a blood pressure, the duration of ROSC is key element not only to the efficacy of the chain of survival but also to assess the success of resuscitation in emergency medical services (EMSs).

Worldwide CPR outcomes vary due to differences in the circumstances of cardiac arrest, availability of equipment, and performance of the CPR team. The influencing factors of CPR outcome at the emergency room (ER) are patient characteristics, early detection, immediate CPR, initial shockable rhythm, duration of CPR of less than 10 minutes and advanced cardiac life support.

In Egypt, There has been scarce studies regarding CPR and studies that measure the success rate of CPR and factors determining its success. This study aims to assess the success rate of CPR in Emergency room and factors predicting successful CPR on adults.

ELIGIBILITY:
Inclusion Criteria:

* Resuscitated at the ER in Al Hussein University Hospital.
* Patients Have experienced cardiac arrest.

Exclusion Criteria:

* Patient arresting and receiving CPR inside hospital's other departments.
* Signs of sure death.
* Patient with Multiple Organ Failure Syndrome (M.O.F syndrome

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
CPR Success Rate | From base line to 20 minutes.
  The rate of CPR defined by the Return of spontaneous circulation(ROSC) rate, Survival to hospital admission rate and survival to hospital discharge rate.

SECONDARY OUTCOMES:
predictors of Return of spontaneous circulation(ROSC) | from base line to 8 hoiurs
  ROSC was defined as a clinical assessment that shows signs of life comprising of a palpable pulse for at least 20 minutes or generating a blood pressure, the duration of ROSC is key element not only to the efficacy of the chain of survival but also to assess the success of resuscitation in emergency medical services

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Mohamed Abdelgaleel, Professor, Study Chair — Al-Azhar University, Faculty of medicine for boys
Locations (1):
- Alhusein Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No